CLINICAL TRIAL: NCT05939856
Title: Lymph Node Dissection Before or After Cystectomy - Pilot Randomized Controlled Trial
Brief Title: Lymph Node Dissection Before or After Cystectomy
Acronym: LBOACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Anna K. Czech, MD, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBOACPUJ
Record Dates: First submitted 2023-06-06; First posted 2023-07-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Muscle-invasive bladder cancer; Radical cystectomy; Lymph node dissection
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Lymph node dissection before bladder resection (Other): Lymph node dissection will be performed before bladder resection during radical cystectomy
  Interventions: Other: Lymph node dissection before bladder resection
- 2 Lymph node dissection after bladder resection (Other): Lymph node dissection will be performed after bladder resection during radical cystectomy
  Interventions: Other: Lymph node dissection after bladder resection

INTERVENTIONS:
Other: Lymph node dissection before bladder resection — Lymph node dissection before bladder resection
  Arms: 1 Lymph node dissection before bladder resection
Other: Lymph node dissection after bladder resection — Lymph node dissection after bladder resection
  Arms: 2 Lymph node dissection after bladder resection

SUMMARY:
The purpose of this study is to compare different ways of performing surgery for bladder cancer. Specifically, the goal is to determine whether it is better to remove the lymph nodes before removing the bladder or after removing the bladder during radical cystectomy.

The study aims to answer two main questions:

* Does the order of surgical steps during radical cystectomy affect the occurrence of complications after surgery?
* Does the order of surgical steps during radical cystectomy impact the duration of the operation and the number of lymph nodes removed?

Participants in the study will be randomly assigned to one of two groups. One group will undergo lymph node removal before bladder resection, while the other group will have lymph node removal after bladder resection during radical cystectomy.

Throughout their hospital stay and for 30 days following the operation, participants will be closely monitored for various factors including operative details, pathology results, and any complications that may arise.

DETAILED DESCRIPTION:
Lymph node dissection (LND) is an integral part of radical cystectomy (RC) for bladder cancer. LND provides important diagnostic and prognostic information, and according to most studies, is associated with therapeutic benefit. The optimal extent and template for LND in bladder cancer remains to be established. Currently, there are no specific recommendations regarding the sequence of lymph nodes removal and bladder resection during radical cystectomy, and the decision is based mainly on individual surgeon preference.

The aim of the LBOAC pilot randomized trial is to evaluate the difference in intraoperative parameters and postoperative outcomes between patients undergoing LND before bladder resection during RC and those undergoing LND after bladder resection during RC.

LBOAC is a pilot randomized controlled trial with two parallel groups. The primary objective of the trial is the comparison of complication rate within 30 postoperative days. Secondary objectives of LBOAC include comparing lymph node yield and operative time between the two groups.

Data for will be collected using electronic case report forms (eCRFs) at baseline and within 30 days after the surgery.

This pilot study is designed to test feasibility of, to support the refinements of the protocol and to aid in sample calculation that can be used for larger scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical cystectomy for bladder cancer in the Department of Urology University Hospital in Krakow

Exclusion Criteria:

* Previous pelvic lymph node dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Early complications rate | Within 30 days after the surgery
  Complications rate within 30 postoperative days

SECONDARY OUTCOMES:
Lymph node yield | When pathology report is available (on average, the pathology report is available within 14 days after the surgery)
  Number of lymph nodes removed
Operative time | At the end of the surgery (after the completion of skin closure and wound dressing)
  Total operative time, bladder resection time, lymph node dissection time

OTHER OUTCOMES:
Intraoperative complications rate | At the end of the surgery (after the completion of skin closure and wound dressing)
  Intraoperative complications rate
Positive surgical margin rate | When pathology report is available (on average, the pathology report is available within 14 days after the surgery)
  Positive surgical margin rate
Ureters clamping time | At the end of the surgery (after the completion of skin closure and wound dressing)
  Ureters clamping time
Postoperative estimated glomerular filtration rate (eGFR) | Within 7 days after the surgery
  eGFR on postoperative day 1 and day 4-7
Complications severity and type | Within 30 days after the surgery
  Severity and type of complications

CONTACTS AND LOCATIONS:
Overall Officials: Anna K. Czech, Principal Investigator — Jagiellonian University
Locations (1):
- Department of Urology, University Hospital, Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No